CLINICAL TRIAL: NCT01022970
Title: A Double Blinded Randomized Placebo-controlled Trial of Intravenous QAX576 in the Treatment of Eosinophilic Esophagitis (EoE)
Brief Title: Efficacy and Safety of QAX576 in Patients With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAX576A2205
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: Esophagitis; Digestive System Diseases; Esophageal disorder; Eosinophilic esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Digestive System Diseases; Esophageal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: QAX576 placebo
- QAX576 (Active Comparator)
  Interventions: Drug: QAX576

INTERVENTIONS:
Drug: QAX576 placebo
  Arms: Placebo
Drug: QAX576
  Arms: QAX576

SUMMARY:
This study is designed to investigate the effects of a 12 week course of intravenous QAX576 6mg/kg every 4 weeks in reducing the number of eosinophils in the esophagus of EoE patients by 75% or greater when compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-50 with symptomatic eosinophilic esophagitis
* Female subjects must be women of non child bearing potential.
* Elimination diet must have been tried.
* Treatment for at least two months prior to enrollment on a protocol pump inhibitor .
* Appropriate contraception must be used by males, (e.g., spermicidal gel plus condom)
* Must be able to communicate well with the investigator, to understand and comply with the requirements of the study.
* Understand and sign the written informed consent.

Exclusion criteria:

* Have received corticosteroids within 3 months before starting the study for any symptoms.
* Any other eosinophilic disorders.
* History of clinical schistosomiasis, or having travelled within the preceding 6 months to an area with endemic schistosomiasis, including but not limited to Southeast and Southwest Asia, South America and Africa. Travel to these areas must not be planned for at least 6 months after the last dose.
* Donation or loss of 400 ml or more of blood within eight (8) weeks prior to initial dosing.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this study is the number of patients (responder) with a reduction of 75% or more in eosinophils per HPF (distal or proximal esophagus) from baseline to week 13. | 13 weeks

SECONDARY OUTCOMES:
To ascertain the effect of QAX576 in the frequency and severity of the symptoms of EoE. | 34 weeks
To investigate the safety and tolerability of QAX576 in patients with EoE. | 34 weeks
To establish the duration of clinical benefit after a 12 week course of therapy. | 34 weeks
PK/PD relationship between blood levels of QAX576 and IL- 13 dependent gene expression in esophageal biopsies and soluble biomarkers, inflammatory and fibrotic markers within esophageal biopsies and activation markers expressed on peripheral | 34 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford Medical Center and Lucile Packard Children's Hospital, Stanford, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Mayo Clinic, Minneota, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oral Alpan, 6210 Old Keene Mill Court,, Springfield, Virginia

REFERENCES:
- [Derived] Rothenberg ME, Wen T, Greenberg A, Alpan O, Enav B, Hirano I, Nadeau K, Kaiser S, Peters T, Perez A, Jones I, Arm JP, Strieter RM, Sabo R, Gunawardena KA. Intravenous anti-IL-13 mAb QAX576 for the treatment of eosinophilic esophagitis. J Allergy Clin Immunol. 2015 Feb;135(2):500-7. doi: 10.1016/j.jaci.2014.07.049. Epub 2014 Sep 13. PMID 25226850
- See also: Results for CQAX576A2205 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8985